CLINICAL TRIAL: NCT03916523
Title: Effect of Sustained Lung Inflation During CPAP in Preterm Neonates With Respiratory Distress Syndrome
Brief Title: Sustained Lung Inflation With CPAP in Preterm Neonates (SI-CPAP)
Acronym: SI-CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada Ibrahim Gad, Professor of Pediatrics, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02072012
Record Dates: First submitted 2019-04-13; First posted 2019-04-16 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: RDS of Prematurity
Keywords: Sustained lung inflation; Lung injury; Delivery room management; CPAP
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Lung Injury | interventions — Continuous Positive Airway Pressure; Respiration, Artificial

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All laboratory testing will be performed by investigators who are not aware of group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Infants in the group receive CPAP for respiratory support in the delivery room. In addition, they receive a total of 15 sustained lung inflations in the first 96 hours of life; 6 in the first day, 3 in the second day, 3 in the third day and 3 in the forth day of life.
  Interventions: Procedure: Sustained lung inflation
- Group B (Experimental): Infants in the group receive CPAP for respiratory support in the delivery room. No sustained lung inflation will be applied.
  Interventions: Procedure: Continuous positive airway pressure (CPAP)
- Group C (Active Comparator): Infants in this group are intubated in the delivery room and supported with mechanical ventilation.
  Interventions: Procedure: Mechanical ventilation

INTERVENTIONS:
Procedure: Sustained lung inflation — Preterm infants will receive a total of 15 sustained lung inflations during the first 4 days of life as follows:
  1. On day 1 of life (a total of 6 sustained lung inflations, 20 cmH2O for 21 seconds each) once at enrollment and then once every 4 hours
  2. On day 2 of life (a total of 3 sustained lung inflations, 15 cmH2O for 21 seconds each) once every 8 hours.
  3. On day 3 of life (a total of 3 sustained lung inflations 10cmH2O for 21 seconds each) once every 8 hours.
  4. On day 4 of life (a total of 3 sustained lung inflations 10cmH2O for 21 seconds each) once every 8 hours.
  Arms: Group A
Procedure: Continuous positive airway pressure (CPAP) — Preterm infants will receive CPAP for respiratory support.
  Other Names: CPAP
  Arms: Group B
Procedure: Mechanical ventilation — Preterm infants in this group will receive mechanical ventilation for respiratory support
  Arms: Group C

SUMMARY:
Neonatal respiratory distress syndrome (RDS) is the most common cause of respiratory failure in the first few days in life. It is characterized by the tendency of alveoli and terminal bronchioles to collapse due to the lack of surfactant. RDS is inversely related to gestational age and remains a dominant clinical problem encountered among preterm infants.

The reduction in tidal volume secondary to alveolar collapse may result in alveolar derecruitment, cyclic opening and closing of atelectatic alveoli and distal small airways leading to inflammation and lung injury). On the other hand, the use of high positive end expiratory pressure (PEEP) may be associated with excessive lung parenchyma strain and unfavorable hemodynamic effects. Therefore, lung recruitment maneuvers have been proposed and used to open collapsed lung while managing with low pressure PEEP. However, the best recruitment maneuver technique is currently unknown.

Proinflammatory cytokines are synthesized by alveolar macrophages, type II pneumocytes and other local pulmonary cells causing inflammation that starts a cascade leading to lung injury. Nevertheless, they are released systemically and can lead to injury of other organs.

This study aims to measure inflammatory cytokines in the serum of premature infants who receive and do not receive sustained lung inflation. The study hypothesis is that, in premature infants supported with CPAP, the use of sustained inflation is associated with decreased inflammatory biomarkers and improved respiratory outcomes.

The study includes infants with gestational age of 28-24 weeks during the first 6 hours of life who will be randomly assigned to either receive (or do not receive) sustained inflations. Serum concentrations of cytokines (IL-6, IL-8, IL-1β and TNF-α) will be measured at enrollment and at 96 hours. The primary outcome of this study will be the change in serum cytokine concentrations after intervention in both groups. Clinical respiratory outcomes will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age between 28 weeks (and 0 days) and 34 weeks (and 6 days)
2. Postnatal age <6 hours
3. Respiratory distress syndrome diagnosed by both clinical findings of subcostal retractions, tachypnea (>70 breaths/min), the need for respiratory support to maintain oxygen saturation > 87% and X-ray findings of RDS
4. Application of early CPAP <6 hours of age
5. Oxygen requirement (FiO2 >30% to maintain preductal saturation 87% - 93%)

Exclusion Criteria:

* Before enrollment: infants will not be considered in the study if any of the following conditions exists: major congenital anomalies, severe hemodynamic instability indicative of early septicemia, use of inotropes, severe metabolic acidemia with base deficit >12 mEq/dl, frequent apnea / bradycardia (6 episodes per day with HR <100 or 2 episodes per day with HR<60 requiring bag-and-mask ventilation), maternal chorioamnionitis (fever >38 degree Celsius with abdominal tenderness) and PPROM >18 hours, and perinatal hypoxia (Apgar score < 6 at 5 minutes)
* After enrollment: infants will be eliminated from the study if the initial blood culture on admission is positive.

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
Serum concentration of cytokines | At 96 hours of life
  IL-6, IL-8, IL-1β, - TNF-α and elastase will be measured in all subjects in group, group B, and group C.

SECONDARY OUTCOMES:
Oxygen requirement | At 96 hours of life
  Fraction of inspired oxygen (FiO2) while on CPAP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Hady H, Shouman B, Aly H. Early weaning from CPAP to high flow nasal cannula in preterm infants is associated with prolonged oxygen requirement: a randomized controlled trial. Early Hum Dev. 2011 Mar;87(3):205-8. doi: 10.1016/j.earlhumdev.2010.12.010. Epub 2011 Jan 26. PMID 21276671
- [Background] Aly H. Ventilation without tracheal intubation. Pediatrics. 2009 Aug;124(2):786-9. doi: 10.1542/peds.2009-0256. Epub 2009 Jul 27. No abstract available. PMID 19651592
- [Background] Attar MA, Donn SM. Mechanisms of ventilator-induced lung injury in premature infants. Semin Neonatol. 2002 Oct;7(5):353-60. doi: 10.1053/siny.2002.0129. PMID 12464497
- [Background] Lista G, Fontana P, Castoldi F, Cavigioli F, Dani C. Does sustained lung inflation at birth improve outcome of preterm infants at risk for respiratory distress syndrome? Neonatology. 2011;99(1):45-50. doi: 10.1159/000298312. Epub 2010 Jul 9. PMID 20616570